CLINICAL TRIAL: NCT04393545
Title: A Comparison of the Effectiveness of Splinting, Exercise and Electrotherapy in the Management of Hallux Valgus: a Randomized Clinical Trial
Brief Title: Efficacy of Splinting, Exercise and Electrotherapy on Hallux Valgus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Bahar Anaforoglu Külünkoglu, ASSOCIATE PROFESSOR, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KA08/143
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Hallux Valgus
Keywords: hallux valgus; Night splint; Exercise; High voltage galvanic stimulation; Radiographic angular degree; Foot-specific health-related quality of life
MeSH Terms: conditions — Hallux Valgus; Motor Activity | interventions — Exercise; Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HV night splint (SP) group (Active Comparator)
  Interventions: Device: hallux valgus night splint
- exercise (EX) group (Active Comparator)
  Interventions: Other: exercise
- high-voltage galvanic stimulation (EL) group (Active Comparator)
  Interventions: Other: Electrotherapy

INTERVENTIONS:
Device: hallux valgus night splint — The HV night splint holds the hallux in abduction in order to provide a correct position. The SP group was given splints consisting of a rigid polyethylene bar along the medial of the hallux, and soft polyform and Velcro fastener parts.
  Arms: HV night splint (SP) group
Other: exercise — The exercises involved strengthening the AbdH (abductor hallucis) and plantar fascia muscles, and stretching the hallux
  Arms: exercise (EX) group
Other: Electrotherapy — Two self-adhesive electrodes were used. One was placed over the medial distal end of the first metatarsal and the other was attached to the motor point of the AbdH (inferior and posterior to the navicular tuberosity).21 The stimulation intensity was increased until a contraction was observed without causing discomfort and pain. Twenty-minute HVPGS was applied in total over three weekly sessions for four weeks.
  Arms: high-voltage galvanic stimulation (EL) group

SUMMARY:
The aim of this study was to investigate the effects of splinting, exercise and electrotherapy on the hallux valgus (HV) angle, and foot-specific health-related quality of life. Sixty women (120 feet) with bilateral HV deformity were randomly assigned to one of three groups - an HV night splint (SP) group, an exercise (EX) group, and a high-voltage galvanic stimulation (EL) group. Angular degrees (hallux interphalangeal, HV, and intermetatarsal angles expressed as angles A, B and C, respectively) were determined before enrollment (t0) and three months after treatment (t2). Foot-specific quality of life was assessed using the Manchester-Oxford Foot Questionnaire (MOFQ) at t0, after one month (t1), and at t2. All groups exhibited significant changes in the A, B, and C angles and outcome measures (p ≤0.001). Decreases in the A and C angles, and MOFQ-Pain subscale scores, were higher in the SP group than in the other two groups (p<0.05). C angle at t2, MOFQ-Walking score at t1 and t2 and MOFQ-Pain subscale score at t1 were lower in the SP group (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of HV confirmed by an orthopedist experienced in foot surgery
* female gender
* bilateral HV deformity
* aged 18-60 years.
* Patients were then selected based on an HV deformity degree of '2' or '3' on the Manchester scale before randomization

Exclusion Criteria:

* Patients with HV deformity degrees less than '2' or more than '3' according to the Manchester scale
* Patients with systemic disease, cognitive or mental disturbance, a history of surgery to the lower extremity, or previous use of any foot splints were excluded.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-02-02 (Actual); Primary Completion 2014-07-07 (Actual); Study Completion 2014-11-03 (Actual)

PRIMARY OUTCOMES:
Manchester Scale | used once before enrollment for the inclusion
  This scale determines the severity of HV and deformity using four foot photographs (0 'no deformity', 1 'mild', 2 'moderate' or 3: 'severe deformity').
change in hallux valgus angle | were taken before enrollment and at three-month follow-up controls
  Antero-posterior radiographs of patients' bilateral feet were taken before treatment and at three-month follow-up controls (in a standing position). HV, intermetatarsal, and hallux interphalangeal angles were measured on the radiographic images. These angles were abbreviated to angles A, B and C respectively.
change in Manchester-Oxford Foot Questionnaire score | were assessed three times: before enrollment, at 1st and 3rd months.
  MOFQ Foot health-related quality of life was evaluated using the MOFQ. This consists of three categories - pain, walking/standing, and social interaction. The MOFQ contains 16 items, each scored on a Likert scale between 0 and 4. Possible scores for each domain range from 0 to 100, with higher scores indicating the most severe conditions

REFERENCES:
- [Derived] Kulunkoglu BA, Akkubak Y, Celik D, Alkan A. A comparison of the effectiveness of splinting, exercise and electrotherapy in women patients with hallux valgus: A randomized clinical trial. Foot (Edinb). 2021 Sep;48:101828. doi: 10.1016/j.foot.2021.101828. Epub 2021 May 25. PMID 34388424